CLINICAL TRIAL: NCT00344747
Title: Multidisciplinary Ambulatory Intervention Program (Dietary Behavioral Physical Activity) in Family of Children and Adolescents With Obesity
Brief Title: Multidisciplinary Ambulatory Intervention Program in Family of Children and Adolescents With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR433806CTIL
Record Dates: First submitted 2006-06-25; First posted 2006-06-27 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Obesity
Keywords: intervention program; diet; physical activity; adolescents; obesity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Diet; Exercise

INTERVENTIONS:
Behavioral: dietary, behavioral, physical activity

SUMMARY:
Obesity has become a pandemic, and it is today's principal neglected public health problem.

Obesity has increased dramatically during the past two decades At adolescence, it is an aggravating issue, because obesity tends to persist in adulthood and the longer its duration, the higher the associated mortality and morbidity. Obesity imposes a heavy health and social burden, and it is widely recognized that treatment is costly. If obesity is not successfully addressed by late adolescence, the likelihood of weight loss in adulthood is as low as 5%. Therefore, prevention is crucial, and children and adolescents should be a priority target.

Treatment of obesity is costly, time consuming, difficult and the results aren't always satisfying On most cases the patients receive dietary advice only (6-10 visits per year). And usually the patients end the treatment early due to lack of results.

The best treatment of children and adolescent obesity is done in highly specialized settings, by a multidisciplinary team. Those programs have a limited number of locations (not always in proximity to the patients' residence), in addition, they are long term treatments and therefore are hard to complete successfully without additional support, Therefore only a limited number of patients can benefit from such programs.

Due to the reasons mentioned above, many families tend not to start the process of treating their obese child, or turn to commercial weight loss programs, or put their children according to their beliefs and diets.

Therefore ambulatory medicine is the ideal setting for the treatment of children and adolescent's obesity, it's also in proximity to the patients' residence, the medical team has a deep knowing of their patients and the possibility for long term maintenance and follow-up.

We propose a trial of obesity treatment by behavior modification program, including parents as agents of change.

ELIGIBILITY:
Inclusion Criteria:Children (6-18 years) with BMI in the 85th to 95th percentile or higher

Exclusion Criteria:Children with chronic diseases treated with chronic medications.

Refuse to participate in to the study

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-09; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
changes in BMI, activity level and Quality of Life questionnaire for the parents and the others children in the family

CONTACTS AND LOCATIONS:
Overall Officials: Gherta Bril, MD, Principal Investigator — BGU
Locations (1):
- Clalit Health Services,, Beersheba, Israel